CLINICAL TRIAL: NCT01360632
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of the Safety and Efficacy of Two Fixed Doses of OPDC-34712 as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder, the Polaris Trial
Brief Title: Study of the Safety and Efficacy of Two Fixed Doses of OPC-34712 as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder (the Polaris Trial)
Acronym: Polaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-10-227
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders
Keywords: OPC-34712; brexpiprazole; Major Depressive Disorder; Adjunctive Treatment
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders | interventions — Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase B (Experimental): Drug: OPC-34712 + ADT
  Drug: Placebo + ADT
  Interventions: Drug: OPC-34712 + ADT; Drug: Placebo + ADT
- Phase A (Placebo Comparator): Drug: Placebo + ADT
  Interventions: Drug: Placebo + ADT

INTERVENTIONS:
Drug: OPC-34712 + ADT — Tablets, Oral, 1 or 3 mg OPC-34712 and FDA Approved Antidepressant Therapy (ADT)
  Arms: Phase B
Drug: Placebo + ADT — Placebo + FDA Approved Antidepressant (ADT)
  Arms: Phase B
Drug: Placebo + ADT — Placebo + FDA Approved Antidepressant (ADT)
  Arms: Phase A

SUMMARY:
To compare the effect of OPC-34712 (brexpiprazole) to the effect of placebo (an inactive substance) as add on treatment to an assigned FDA approved antidepressant treatment (ADT) in patients with Major Depressive Disorder who demonstrate an incomplete response to a prospective trial of the same assigned FDA approved ADT

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age, with diagnosis of major depressive disorder, as defined by DSM-IV-TR criteria
* The current depressive episode must be equal to or greater than 8 weeks in duration
* Subjects must report a history for the current depressive episode of an inadequate response to no more than three adequate antidepressant treatments

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug
* Subjects who report an inadequate response to more than three adequate trials of antidepressant treatments during current depressive episode at a therapeutic dose for an adequate duration
* Subjects with a current Axis I (DSM-IV-TR) diagnosis of: Delirium, dementia, amnestic or other cognitive disorder, Schizophrenia, schizoaffective disorder, or other psychotic disorder, Bipolar I or II disorder
* Subjects with a clinically significant current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1539 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (52):
  - Research Site, Birmingham, Alabama
  - Research Site, Costa Mesa, California
  - Research Site, Glendale, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Temecula, California
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Lafayette, Indiana
  - Research Site, Owensboro, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Haverhill, Massachusetts
  - Research Site, Weymouth, Massachusetts
  - Research Site, Rochester Hills, Michigan
  - Research Site, Creve Coeur, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Salem, Oregon
  - Research Site, Norristown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Witchita Falls, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Herndon, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Spokane, Washington
  - Research Site, Brown Deer, Wisconsin
  - Research Site, Middleton, Wisconsin
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec
- Germany (4):
  - Research Site, Würzburg, Bavaria
  - Research Site, Stralsund, Mecklenburg-Vorpommern
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Achim
- Hungary (3):
  - Research Site, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Research Site, Budapest
  - Research Site, Győr
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Lasi
  - Research Site, Târgu Mureş
- Russia (3):
  - Research Site, Moscow
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
- Ukraine (4):
  - Research Site, Chenigiv
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Poltava

REFERENCES:
- [Derived] Kapadia S, Zhang Z, Ardic F, Patel M, Thase ME, Papakostas GI. Adjunctive brexpiprazole in patients with major depressive disorder who show minimal or partial response to antidepressant treatment: post hoc analysis of randomized controlled trials. Int J Neuropsychopharmacol. 2025 Oct 1;28(10):pyaf074. doi: 10.1093/ijnp/pyaf074. PMID 41055581
- [Derived] Ardic F, Zhang Z, Hogan M. Effects of adjunctive brexpiprazole in patients with major depressive disorder and sleep disturbance: a post hoc analysis of three randomized trials. Front Psychiatry. 2025 Aug 7;16:1618176. doi: 10.3389/fpsyt.2025.1618176. eCollection 2025. PMID 40852147
- [Derived] Kapadia S, Zhang Z, Csoboth C, Patel M, Thase ME, Papakostas GI. Adjunctive brexpiprazole in patients with unresolved symptoms of depression on antidepressant treatment who are early in the disease course: post hoc analysis of randomized controlled trials. Int J Neuropsychopharmacol. 2025 Aug 1;28(8):pyaf050. doi: 10.1093/ijnp/pyaf050. PMID 40607746
- [Derived] McIntyre RS, Bubolic S, Zhang Z, MacKenzie EM, Therrien F, Miguelez M, Boucher M. Effects of Adjunctive Brexpiprazole on Individual Depressive Symptoms and Functioning in Patients With Major Depressive Disorder and Anxious Distress: Post Hoc Analysis of Three Placebo-Controlled Studies. J Clin Psychopharmacol. 2024 Mar-Apr 01;44(2):133-140. doi: 10.1097/JCP.0000000000001825. PMID 38421922
- [Derived] Newcomer JW, Meehan SR, Chen D, Brubaker M, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Prediabetes Treated With Adjunctive Brexpiprazole for Major Depressive Disorder: Pooled Analysis of Short- and Long-Term Clinical Studies. J Clin Psychiatry. 2023 Aug 28;84(5):23m14786. doi: 10.4088/JCP.23m14786. PMID 37656180
- [Derived] McIntyre RS, Therrien F, Ismail Z, Meehan SR, Miguelez M, Larsen KG, Chen D, MacKenzie EM, Thase ME. Effects of adjunctive brexpiprazole on patient life engagement in major depressive disorder: Post hoc analysis of Inventory of Depressive Symptomatology Self-Report data. J Psychiatr Res. 2023 Jun;162:71-78. doi: 10.1016/j.jpsychires.2023.04.012. Epub 2023 Apr 12. PMID 37099968
- [Derived] Newcomer JW, Eriksson H, Zhang P, Meehan SR, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Major Depressive Disorder Treated With Adjunctive Brexpiprazole: Pooled Analysis of Phase 3 Clinical Studies. J Clin Psychiatry. 2019 Oct 1;80(6):18m12680. doi: 10.4088/JCP.18m12680. PMID 31577867
- [Derived] Hobart M, Zhang P, Weiss C, Meehan SR, Eriksson H. Adjunctive Brexpiprazole and Functioning in Major Depressive Disorder: A Pooled Analysis of Six Randomized Studies Using the Sheehan Disability Scale. Int J Neuropsychopharmacol. 2019 Mar 1;22(3):173-179. doi: 10.1093/ijnp/pyy095. PMID 30508090
- [Derived] McIntyre RS, Weiller E, Zhang P, Weiss C. Brexpiprazole as adjunctive treatment of major depressive disorder with anxious distress: Results from a post-hoc analysis of two randomised controlled trials. J Affect Disord. 2016 Sep 1;201:116-23. doi: 10.1016/j.jad.2016.05.013. Epub 2016 May 12. PMID 27208498
- [Derived] Thase ME, Youakim JM, Skuban A, Hobart M, Zhang P, McQuade RD, Nyilas M, Carson WH, Sanchez R, Eriksson H. Adjunctive brexpiprazole 1 and 3 mg for patients with major depressive disorder following inadequate response to antidepressants: a phase 3, randomized, double-blind study. J Clin Psychiatry. 2015 Sep;76(9):1232-40. doi: 10.4088/JCP.14m09689. PMID 26301771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 1539 participants at 92 trial sites in 7 countries. United States, Germany, Ukraine, Russia, Hungary, Canada, and Romania.
Pre-assignment Details: The study consisted of a 7 to 28-day Screening period, an 8-Week single-blind placebo + ADT prospective Phase-A, a 6-Week double-blind randomization Phase-B or single-blind Phase A+ and a Follow-up of 30 (+2) days after the last dose of study medication.
Groups:
- Single-blind Placebo + ADT: In Phase A, participants were administered placebo as an adjunctive therapy to an open label ADT for 8 weeks.
- Brexpiprazole (1mg) + ADT: Participants were administered brexpiprazole of [1mg (milligram)] as an adjunctive therapy to an assigned open-label ADT (anti-depressant therapy).
- Brexpiprazole (3mg) + ADT: Participants were administered brexpiprazole of 3mg as an adjunctive therapy to an assigned open-label ADT.
- Double-blind Placebo + ADT: In phase B, participants were administered placebo as an adjunctive therapy to an open label ADT for 6 weeks.
- Phase A+ Placebo + ADT: Participants who did not meet criteria for randomization and a follow-up of 30 (+2) days after the last dose of study medication were in Phase A+
Period: Phase A (8 Weeks)
Arm/Group | Single-blind Placebo + ADT | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Double-blind Placebo + ADT | Phase A+ Placebo + ADT
Started | 1532 (A total of 1539 participants were enrolled, 7 discontinued before taking any sponsor-provided ADT) | 0 (These participants were from the randomized sample.) | 0 (These participants were from the randomized sample.) | 0 (These participants were from the randomized sample.) | 0
Completed | 1277 | 0 | 0 | 0 | 0
Not Completed | 255 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 27 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 60 | 0 | 0 | 0 | 0
Not completed — Met Withdrawal Criteria | 45 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 10 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 74 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 39 | 0 | 0 | 0 | 0
Period: Phase B (6 Weeks)
Arm/Group | Single-blind Placebo + ADT | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Double-blind Placebo + ADT | Phase A+ Placebo + ADT
Started | 0 | 226 (These participants were from the randomized sample.) | 230 (These participants were from the randomized sample.) | 221 (These participants were from the randomized sample.) | 0
Completed | 0 | 216 | 210 | 208 | 0
Not Completed | 0 | 10 | 20 | 13 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 9 | 3 | 0
Not completed — Met Withdrawal Criteria | 0 | 0 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 4 | 7 | 0
Not completed — Protocol Deviation | 0 | 1 | 4 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Period: Phase A+
Arm/Group | Single-blind Placebo + ADT | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Double-blind Placebo + ADT | Phase A+ Placebo + ADT
Started | 0 | 0 | 0 | 0 | 600
Completed | 0 | 0 | 0 | 0 | 575
Not Completed | 0 | 0 | 0 | 0 | 25
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Met Withdrawal Criteria | 0 | 0 | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 8
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole (1mg + ADT): Participants were administered brexpiprazole of 1mg as an adjunctive therapy to an assigned open-label ADT.
- Brexpiprazole (3mg + ADT): Participants were administered brexpiprazole of 3mg as an adjunctive therapy to an assigned open-label ADT.
- Placebo + ADT: Participants were administered placebo as an adjunctive therapy to an open label ADT.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole (1mg + ADT) | Brexpiprazole (3mg + ADT) | Placebo + ADT | Total
Number analyzed (Participants) | 226 | 230 | 221 | 677
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (11.6) | 44.5 (11.2) | 46.6 (11.0) | 45.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 156 | 146 | 460
  Male | 68 | 74 | 75 | 217

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From the End of Phase A (Week 8 Visit) to Phase B (Week 14 Visit) in the Montgomery-Asberg Depression Rating Scale for the Efficacy Sample Set
Description: The MADRS was utilized as the primary efficacy assessment of a participant's level of depression. The MADRS consisted of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS total score were to be unevaluable if less than 8 of the 10 items were recorded. If 8 or 9 of the 10 items were recorded, the MADRS total score was the mean of the recorded items multiplied by 10 and then rounded of to the first decimal place. The MADRS Total Score is the sum of ratings for all 10 items. The possible total scores are from 0 to 60, with higher values indicating worse outcome.
Time Frame: Baseline and Week 14
Population: The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole (1mg) + ADT: Participants were administered brexpiprazole 1mg/day as an adjunctive therapy to an assigned open-label ADT.
- Brexpiprazole (3mg) + ADT: Participants were administered brexpiprazole 3mg/day as an adjunctive therapy to an assigned open-label ADT.
- Placebo + ADT: Participants were administered placebo daily as an adjunctive therapy to an open label ADT.
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale | -7.65 (0.5) | -7.98 (0.51) | -6.45 (0.51)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; The primary analysis was performed on the Efficacy Sample by fitting a Mixed Model Repeated Measures (MMRM) analysis with an unstructured variance covariance structure in which the change from the end of Phase A (Week 8) in MADRS Total Score (at Weeks 9 to 14) was the dependent variable. The model included fixed class effect terms for treatment, trial site, visit week, and an interaction term of treatment by visit week; Test type: Superiority or Other; p = 0.0925, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-2.58 to 0.2]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; The primary analysis was performed on the Efficacy Sample by fitting a MMRM analysis with an unstructured variance covariance structure in which the change from the end of Phase A (Week 8) in MADRS Total Score (at Weeks 9 to 14) was the dependent variable. The model included fixed class effect terms for treatment, trial site, visit week, and an interaction term of treatment by visit week; Test type: Superiority or Other; p = 0.0327, Mixed Models Analysis; MMRM method was used with trial site, treatment group, visit, treatment group-by-visit and Baseline-by-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.52, 95% CI 2-sided [-2.92 to -0.13]

2. Primary Outcome: Mean Change in MADRS Total Score From Baseline End of Week 8 to Week 14 for the Efficacy Sample Per Final Protocol
Description: as for outcome 1
Time Frame: Baseline and Week 14
Population: Analysis was based on all participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Units on a scale | -7.64 (0.52) | -8.29 (0.53) | 6.33 (0.53)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0737, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-2.73 to 0.13]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0079, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-3.39 to -0.51]

3. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) in MADRS Total Score for Every Study Week Visit in Phase B Other Than Week 14 Visit for the Efficacy Sample Set
Description: as for outcome 1
Time Frame: Week 8, 9, 10, 11, 12, and 13
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale
  Week 9 | -3.25 (0.3) | -2.53 (0.3) | -2.19 (0.31)
  Week 10 | -5.34 (0.38) | -4.8 (0.38) | -3.91 (0.39)
  Week 11 | -6.25 (0.41) | -5.56 (0.41) | -4.85 (0.41)
  Week 12 | -7.08 (0.43) | -6.8 (0.44) | -5.52 (0.44)
  Week 13 | -7.55 (0.46) | -7.73 (0.46) | -6.04 (0.47)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis at Week 9. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0096, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-1.86 to -0.26]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4137, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.14 to 0.47]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis at Week 10. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-2.47 to -0.4]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.0914, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-1.93 to 0.14]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis at Week 11. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0139, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-2.5 to -0.28]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.2097, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.82 to 0.4]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis at Week 12. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0099, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-2.75 to -0.38]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-2.48 to -0.1]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis at Week 13. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0177, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-2.8 to -0.27]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.0085, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-2.98 to -0.44]

4. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) in MADRS Total Score for Every Study Week Visit in Phase B Other Than Week 14 Visit for the Efficacy Sample Per Final Protocol
Description: as for outcome 1
Time Frame: Week 8, 9, 10, 11, 12, and 13
Population: All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Units on a scale
  Week 9 | -3.09 (0.31) | -2.6 (0.31) | -2.18 (0.32)
  Week 10 | -5.12 (0.39) | -4.92 (0.39) | -3.95 (0.4)
  Week 11 | -6.22 (0.42) | -5.76 (0.43) | -4.86 (0.43)
  Week 12 | -7.09 (0.45) | -7.11 (0.45) | -5.48 (0.46)
  Week 13 | -7.56 (0.47) | -8.05 (0.48) | -5.93 (0.49)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 9. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0286, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.74 to -0.1]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 9. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.3173, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.24 to 0.4]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 10. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0313, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-2.23 to -0.11]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 10. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0732, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-2.04 to 0.09]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 11. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0206, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-2.51 to -0.21]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 11. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.1233, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-2.06 to 0.25]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 12. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0097, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-2.84 to -0.39]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 12. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0092, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-2.86 to -0.41]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 13. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0139, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-2.94 to -0.33]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 13. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -2.12, 95% CI 2-sided [-3.42 to -0.81]

5. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Sheehan Disability Scale (SDS) Mean Scores for the Efficacy Sample Set
Description: The SDS was a self-rated instrument used to measure the effect of the participants symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores ranged from 0 through 10. The number most representative of how much each area was disrupted by symptoms was marked along the line from 0= not at all to 10= extremely. For the work/school item, no response was to be entered if the participant did not work or go to school for reasons unrelated to the disorder and a response therefore not being applicable. The Mean SDS score were calculated over the three item scores. All three item scores were needed to be available with the exception of the work/school item score when this item was not applicable.
Time Frame: Week 11 and Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale
  Week 11 | -1.13 (0.13) | -0.67 (0.13) | -0.58 (0.11)
  Week 14 | -1.33 (0.14) | -1.21 (0.13) | -0.84 (0.13)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 11. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis — MMRM method was used with trial site, treatment group, visit, treatment group-by-visit and Baseline-by-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.87 to -0.23]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 11. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.5792, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.41 to 0.23]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 14. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0091, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.87 to -0.12]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.0474, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.73 to 0]

6. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in SDS Mean Scores for the Efficacy Sample Per Final Protocol
Description: The SDS was a self-rated instrument used to measure the effect of the participants symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores ranged from 0 through 10. The number most representative of how much each area was disrupted by symptoms was marked along the line from 0= not at all, to 10= extremely. For the work/school item, no response was to be entered if the participant did not work or go to school for reasons unrelated to the disorder and a response therefore not being applicable. The Mean SDS score were calculated over the three item scores. All three item scores were needed to be available with the exception of the work/school item score when this item was not applicable.
Time Frame: Week 11 and Week 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Units on a scale
  Week 11 | -1.11 (0.13) | -0.74 (0.13) | -0.53 (0.14)
  Week 14 | -1.27 (0.15) | -1.26 (0.15) | -0.78 (0.15)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.94 to -0.22]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.2627, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.56 to 0.15]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 14. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0158, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.89 to -0.09]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 14. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3; Test type: Superiority or Other; p = 0.0191, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.88 to -0.08]

7. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) in SDS Item Scores for the Efficacy Sample Set
Description: The SDS is a self-rated instrument used to measure the effect of the patient's symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores range from 0 through 10. The number most representative of how much each area was disrupted by symptoms is marked along the line from 0 = not at all, to 10 = extremely. For the work/school item, no response was to be entered if the patient did not work or go to school for reasons unrelated to the disorder and a response therefore not being applicable. The Mean SDS Score will be calculated over the three item scores. All three item scores need to be available with the exception of the work/school item score when this item is not applicable.
Time Frame: Week 11 and Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale
  Work/school: Week 11 | -1.00 (0.16) | -0.18 (0.18) | -0.55 (0.15)
  Work/school: Week 14 | -1.16 (0.17) | -0.91 (0.18) | -0.73 (0.17)
  Social life: Week 11 | -1.13 (0.14) | -0.76 (0.14) | -0.72 (0.14)
  Social life: Week 14 | -1.39 (0.15) | -1.31 (0.15) | -0.91 (0.15)
  Family life: Week 11 | -1.14 (0.14) | -0.74 (0.14) | -0.51 (0.12)
  Family life: Week 14 | -1.35 (0.15) | -1.28 (0.16) | -0.80 (0.15)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; For Item: Work/School: Week 11; Test type: Superiority or Other; p = 0.0377, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.88 to -0.03]
Statistical Analysis 2: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; For Item: Work/School: Week 14; Test type: Superiority or Other; p = 0.0741, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.91 to 0.04] — -0.43
Statistical Analysis 3: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; For Item: Work/School: Week 11; Test type: Superiority or Other; p = 0.0966, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.07 to 0.81]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; For Item: Work/School: Week 14; Test type: Superiority or Other; p = 0.4774, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.66 to 0.31]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Social life: Week 11; Test type: Superiority or Other; p = 0.0263, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.76 to -0.05]
Statistical Analysis 6: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Social life: Week 14; Test type: Superiority or Other; p = 0.0214, Mixed Models Analysis; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.89 to -0.07]
Statistical Analysis 7: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Social life: Week 11; Test type: Superiority or Other; p = 0.8281, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.40 to 0.32]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Social life: Week 14; Test type: Superiority or Other; p = 0.0540, Mixed Models Analysis; Mean Difference (Net) = -0.40, 95% CI 2-sided [-0.80 to 0.01]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Family life: Week 11; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Net) = -0.63, 95% CI 2-sided [-0.99 to -0.26]
Statistical Analysis 10: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Family life: Week 14; Test type: Superiority or Other; p = 0.0093, Mixed Models Analysis; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.97 to -0.14]
Statistical Analysis 11: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Family life: Week 11; Test type: Superiority or Other; p = 0.2182, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.59 to 0.14]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Family life: Week 14; Test type: Superiority or Other; p = 0.0256, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.90 to -0.06]

8. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) in SDS Item Scores for the Efficacy Sample Set Per Final Protocol
Description: as for outcome 7
Time Frame: Week 11 and Week 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Units on a scale
  Work/school: Week 11 | -1.01 (0.18) | -0.20 (0.20) | -0.48 (0.19)
  Work/school: Week 14 | -1.11 (0.20) | -0.93 (0.21) | -0.65 (0.20)
  Social life: Week 11 | -1.11 (0.15) | -0.82 (0.15) | -0.68 (0.15)
  Social life: Week 14 | -1.34 (0.16) | -1.37 (0.16) | -0.88 (0.17)
  Family life: Week 11 | -1.17 (0.14) | -0.89 (0.15) | -0.54 (0.15)
  Family life: Week 14 | -1.32 (0.16) | -1.39 (0.16) | -0.81 (0.16)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT; Work/school: Week 11; Test type: Superiority or Other; p = 0.0341, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.01 to -0.04]
Statistical Analysis 2: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; School/work: Week 14; Test type: Superiority or Other; p = 0.0816, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.99 to 0.06]
Statistical Analysis 3: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Work/school: Week 11; Test type: Superiority or Other; p = 0.2561, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.21 to 0.78]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Work/school: Week 14; Test type: Superiority or Other; p = 0.2952, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.82 to 0.25]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Social life: Week 11; Test type: Superiority or Other; p = 0.0331, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.82 to -0.03]
Statistical Analysis 6: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Social life: Week 14; Test type: Superiority or Other; p = 0.0352, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.90 to -0.03]
Statistical Analysis 7: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Social life: Week 11; Test type: Superiority or Other; p = 0.4860, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.54 to 0.25]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Social life: Week 14; Test type: Superiority or Other; p = 0.0282, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.93 to -0.05]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Family life: Week 11; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.01 to -0.24]
Statistical Analysis 10: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Family life: Week 14; Test type: Superiority or Other; p = 0.0186, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.94 to -0.09]
Statistical Analysis 11: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Family life: Week 11; Test type: Superiority or Other; p = 0.0824, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.73 to 0.04]
Statistical Analysis 12: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Family life: Week 14; Test type: Superiority or Other; p = 0.0077, Mixed Models Analysis — MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-1.02 to -0.16]

9. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to Phase B by Study Week in Clinical Global Impression Severity of Illness (CGI-S) for the Efficacy Sample Set
Description: The severity of illness for each participant was rated using the CGI-S. To perform this assessment, the study physician had to answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Weeks 8, 9, 10, 11, 12,13 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale
  Week 9 | -0.25 (0.03) | -0.22 (0.03) | -0.16 (0.03)
  Week 10 | -0.52 (0.05) | -0.46 (0.05) | -0.31 (0.05)
  Week 11 | -0.64 (0.05) | -0.51 (0.05) | -0.44 (0.05)
  Week 12 | -0.73 (0.05) | -0.72 (0.05) | -0.59 (0.05)
  Week 13 | -0.78 (0.06) | -0.77 (0.06) | -0.66 (0.06)
  Week 14 | -0.86 (0.06) | -0.9 (0.06) | -0.75 (0.06)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 9. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0436, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.18 to 0]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 9. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = -0.06, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.15 to 0.03]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 10. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.34 to -0.08]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 10. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0266, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.27 to -0.02]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.33 to -0.07]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.3053, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.2 to 0.06]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 12. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0541, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.29 to 0]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 12. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0912, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.28 to 0.02]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 13. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.1553, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.28 to 0.04]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 13. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.1855, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.27 to 0.05]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.2015, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.28 to 0.06]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 14. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B; Test type: Superiority or Other; p = 0.0852, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.32 to 0.02]

10. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to Phase B by Study Week in Clinical CGI-S for the Efficacy Sample Per Final Protocol
Description: as for outcome 9
Time Frame: Weeks 8, 9, 10, 11, 12, 13, and 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Units on a scale
  Week 9 | -0.24 (0.03) | -0.23 (0.03) | -0.16 (0.03)
  Week 10 | -0.5 (0.05) | -0.47 (0.05) | -0.33 (0.05)
  Week 11 | -0.64 (0.05) | -0.53 (0.05) | -0.45 (0.05)
  Week 12 | -0.73 (0.06) | -0.74 (0.06) | -0.58 (0.06)
  Week 13 | -0.77 (0.06) | -0.8 (0.06) | -0.64 (0.06)
  Week 14 | -0.87 (0.06) | -0.92 (0.06) | -0.72 (0.06)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0817, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Median Difference (Final Values) = -0.08, 95% CI 2-sided [-0.17 to 0.01]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.1406, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.16 to 0.02]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.29 to -0.04]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.0287, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.27 to -0.02]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.0071, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.32 to -0.05]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.2503, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.22 to -0.06]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.0539, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.3 to 0]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.0398, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.31 to -0.01]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.1168, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.3 to 0.03]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.0621, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.32 to 0.01]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.089, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.32 to 0.02]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0213, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.38 to -0.03]

11. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) for Every Study Week Visit in Phase B in Inventory of Depressive Symptomatology (Self-Report) IDS-SR Total Score for the Efficacy Sample Set
Description: IDS-SR was a 30-item self-report measured to assess core diagnostic depressive symptoms and atypical and melancholic symptom features of major depressive disorders. The IDS-SR consists of 30 items, all rated on a 0 to 3 scale with 0 being the "best" rating and 3 being the "worst" rating. Besides item 9, two sub-items 9A and 9B exist, with possible scores of 1, 2 or 3 for item 9A, and 0 or 1 for item 9B. The scores for these two sub-items were not included in the calculation of the total score. The IDS-SR Total Score was the sum of ratings of 28 item scores. The possible IDSSR Total Score ranged from 0 to 84. The IDS-SR Total Score was un-evaluable if less than 23 of the 28 items were recorded. If the number of items recorded was at least 23 and at most 27, the IDS-SR Total Score was the mean of the recorded items multiplied by 28, and was then rounded off to the first decimal place.
Time Frame: Weeks 8, 9, 10, 11, 12, 13, and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale
  Week 9 | -3.58 (0.41) | -2.68 (0.42) | -2.31 (0.42)
  Week 10 | -4.97 (0.49) | -4.00 (0.5) | -3.11 (0.5)
  Week 11 | -5.83 (0.56) | -4.15 (0.56) | -3.74 (0.57)
  Week 12 | -6.33 (0.59) | -5.77 (0.59) | -4.43 (0.6)
  Week 13 | -6.96 (0.63) | -6.62 (0.63) | -5.66 (0.64)
  Week 14 | -7.02 (0.66) | -6.94 (0.66) | -5.42 (0.67)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.37 to -0.18]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.5081, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.47 to 0.73]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-3.2 to -0.53]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 4]; Test type: Superiority or Other; p = 0.1898, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-2.23 to 0.44]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0074, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-3.62 to -0.56]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.5935, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.95 to 1.11]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.0211, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.52 to -0.29]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 8]; Test type: Superiority or Other; p = 0.1031, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.96 to 0.27]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 9]; Test type: Superiority or Other; p = 0.1366, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.1366, 95% CI 2-sided [-3.02 to 0.41]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 10]; Test type: Superiority or Other; p = 0.2709, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-2.68 to 0.75]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.0812, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.4 to 0.2]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 9, analysis 12]; Test type: Superiority or Other; p = 0.1001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.52, 95% CI 2-sided [-3.33 to 0.29]

12. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) for Every Study Week Visit in Phase B in IDS-SR Total Score for the Efficacy Sample Per Final Protocol
Description: The IDS-SR was a 30-item self-report measured to assess core diagnostic depressive symptoms as well as atypical and melancholic symptom features of major depressive disorders. The IDS-SR consists of 30 items, all rated on a 0 to 3 scale with 0 being the "best" rating and 3 being the "worst" rating. Besides item 9, two sub-items 9A and 9B exist, with possible scores of 1, 2 or 3 for item 9A, and 0 or 1 for item 9B. The scores for these two sub-items were not included in the calculation of the total score. The IDSSR Total Score was the sum of ratings of 28 item scores. The possible IDSSR Total Score ranged from 0 to 84. The IDS-SR Total Score was un-evaluable if less than 23 of the 28 items were recorded. If the number of items recorded was at least 23 and at most 27, the IDS-SR Total Score was the mean of the recorded items multiplied by 28, and was then rounded off to the first decimal place.
Time Frame: Weeks 8, 9, 10, 11, 12, 13, and 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Units on a scale
  Week 9 | -3.27 (0.42) | -2.65 (0.42) | -2.15 (0.43)
  Week 10 | -4.7 (0.51) | -4.13 (0.51) | -2.94 (0.52)
  Week 11 | -5.77 (0.57) | -4.29 (0.58) | -3.46 (0.59)
  Week 12 | -6.33 (0.61) | -6.05 (0.61) | -4.18 (0.63)
  Week 13 | -6.88 (0.64) | -6.97 (0.64) | -5.25 (0.66)
  Week 14 | -6.97 (0.67) | -7.2 (0.68) | -5.07 (0.69)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0496, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-2.24 to 0]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.387, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.61 to 0.63]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.0125, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-3.13 to -0.38]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.0898, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-2.57 to 0.19]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -2.31, 95% CI 2-sided [-3.88 to -0.74]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.301, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.4 to 0.74]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.0118, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-3.82 to -0.48]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.0287, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.87, 95% CI 2-sided [-3.54 to -0.19]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.0686, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-3.39 to 0.12]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-3.47 to 0.04]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.0448, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.75 to -0.04]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.0251, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-3.98 to -0.27]

13. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) Hamilton Depression Scale 17 Item Version (HAM)-D17 Total Score for the Efficacy Sample Set
Description: The HAM-D17 was utilized as a secondary assessment of a participants level of depression. The HAM-D (17-Item) consisted of 17 items. Eight items were rated on a 0 to 2 scale (items 4, 5, 6, 12, 13, 14, 16 and 17), while nine items (items 1, 2, 3, 7, 8, 9, 10, 11, and 15) were rated on a 0 to 4 scale (twice the weight of the other items). For all of these items, 0 was the "best" rating and the highest score (2 or 4) was the "worst" rating. The possible total scores were from 0 to 52, with higher scores indicating more severe depression.
Time Frame: Baseline and Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 222 | 220 | 213
Units on a scale | -5.47 (0.36) | -6.14 (0.36) | -4.8 (0.37)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 14. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The last observation carried forward (LOCF) method was used to impute missing data; Test type: Superiority or Other; p = 0.1732, ANCOVA; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.63 to 0.29]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 14. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The last observation carried forward (LOCF) method was used to impute missing data; Test type: Superiority or Other; p = 0.0066, ANCOVA; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.31 to -0.37]

14. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in HAM-D17 Total Score for the Efficacy Sample Set Per Final Protocol
Description: The HAM-D17 was utilized as a secondary assessment of a participants level of depression. The HAM-D (17-Item) consisted of 17 items. Eight items were rated on a 0 to 2 scale (items 4, 5, 6, 12, 13, 14, 16 and 17), while nine items (items 1, 2, 3, 7, 8, 9, 10, 11, and 15) were rated on a 0 to 4 scale (twice the weight of the other items). For all of these items, 0 was the "best" rating and the highest score (2 or 4) was the "worst" rating. The possible total scores were from 0 to 52, with higher score indicating more severe depression.
Time Frame: Baseline and Week 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 208 | 207 | 198
Units on a scale | -5.36 (0.37) | -6.26 (0.38) | -4.57 (0.39)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 14. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.1226, ANCOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.78 to 0.21]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 14. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-2.69 to -0.68]

15. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in Hamilton Anxiety Rating Scale (HAM-A) Total Score for the Efficacy Sample Set
Description: The HAM-A is utilized for the evaluation of anxiety symptoms. The HAM-A consists of 14 items. Each item is rated on a 0 to 4 scale. For all of these items, 0 is the "best" rating and 4 is the "worst" rating. If no item scores are missing, then the HAM-A total score is the sum of all 14 item scores. The possible total scores are from 0 to 56, with higher scores indicating worse anxiety symptoms.
Time Frame: Baseline and Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 220 | 216 | 210
Units on a scale | -3.43 (0.31) | -3.89 (0.31) | -3.33 (0.32)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 14. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.8164, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.93 to 0.73]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 14. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.1939, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.39 to 0.28]

16. Secondary Outcome: Mean Change From End of Phase A (Week 8 Visit) to End of Phase B (Week 14 Visit) in HAM-A Total for the Efficacy Sample Per Final Protocol
Description: The HAM-A is utilized for the evaluation of anxiety symptoms. The HAM-A consists of 14 items. Each item is rated on a 0 to 4 scale. For all of these items, 0 is the "best" rating and 4 is the "worst" rating. If no item scores are missing, then the HAM-A total score is the sum of all 14 item scores. The possible total scores are from 0 to 56, with higher score indicating worse anxiety symptoms.
Time Frame: Baseline and Week 14
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 206 | 204 | 195
Units on a scale | -3.35 (0.32) | -3.96 (0.33) | -3.07 (0.33)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.5192, ANCOVA; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.14 to 0.57]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.0443, ANCOVA; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.75 to -0.02]

17. Secondary Outcome: Mean CGI-I Score at Each Trial Week Visit in Phase B for the Efficacy Sample Set
Description: The efficacy of study medication was rated for each participant using the CGI-I. The study physician would rate the participant's total improvement whether or not it is due entirely to drug treatment.
  Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Week 8 to Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale
  Week 9 | 3.36 (0.68) | 3.4 (0.75) | 3.51 (0.67)
  Week 10 | 3.08 (0.85) | 3.09 (0.85) | 3.34 (0.85)
  Week 11 | 2.91 (0.82) | 2.99 (0.89) | 3.17 (0.88)
  Week 12 | 2.78 (0.87) | 2.81 (0.95) | 3.02 (0.95)
  Week 13 | 2.72 (0.87) | 2.73 (1.01) | 2.97 (1.00)
  Week 14 | 2.69 (0.89) | 2.66 (1.1) | 2.85 (1.01)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 9. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0248, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from Cochran-Mantel-Haenszel (CMH) row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.26 to -0.02]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 9. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.1334, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean scores statistics controlling for study center; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.22 to 0.03]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 10. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.42 to -0.11]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 10. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean scores statistics controlling for study center; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.38 to -0.09]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 11. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.42 to -0.11]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 11. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0254, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.34 to -0.02]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 12. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0035, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.41 to -0.08]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 12. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0152, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.39 to -0.04]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 13. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.42 to -0.08]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 13. The Efficacy Sample Set included all participants who had received at least one dose of study treatment and had both an end of Phase A (Week 8) value and at least 1 post randomization efficacy evaluation for MADRS Total Score in Phase B. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.42 to -0.05]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0755, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.33 to 0.02]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.0527, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.39 to 0]

18. Secondary Outcome: Mean CGI-I Score at Each Trial Week Visit in Phase B for the Efficacy Sample Per Final Protocol
Description: as for outcome 17
Time Frame: Weeks 8, 9, 10, 11, 12, 13, and 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Units on a scale
  Week 9 | 3.39 (0.65) | 3.42 (0.74) | 3.54 (0.65)
  Week 10 | 3.1 (0.82) | 3.08 (0.84) | 3.35 (0.84)
  Week 11 | 2.93 (0.8) | 2.99 (0.89) | 3.19 (0.86)
  Week 12 | 2.8 (0.86) | 2.81 (0.94) | 3.06 (0.94)
  Week 13 | 2.75 (0.86) | 2.72 (1) | 3.01 (0.96)
  Week 14 | 2.71 (0.88) | 2.65 (1.09) | 2.9 (0.99)
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 9. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0275, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.26 to -0.01]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 9. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.1583, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.22 to 0.04]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 10. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.41 to -0.09]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 10. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0018, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.4 to -0.09]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 11. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.43 to -0.11]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 11. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0235, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.36 to -0.03]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 12. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.44 to -0.10]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 12. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0111, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.42 to -0.05]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 13. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0030, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.44 to -0.09]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 13. All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.0046, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.47 to -0.09]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0237, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.39 to -0.03]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.0171, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.45 to -0.04]

19. Secondary Outcome: Percentage of Participants With a MADRS Response During Phase B Relative to the End of Phase A (Week 8 Visit) for the Efficacy Sample Set
Description: MADRS response was defined as >=50 percent reduction in MADRS Total Score from end of Phase A (Week 8). The MADRS was utilized as an efficacy assessment of a participant's level of depression. The MADRS consisted of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS total score were to be unevaluable if less than 8 of the 10 items were recorded. If 8 or 9 of the 10 items were recorded, the MADRS total score was the mean of the recorded items multiplied by 10 and then rounded of to the first decimal place. The MADRS Total Score is the sum of ratings for all 10 items. The possible total scores are from 0 to 60, with higher values indicating worse outcome.
Time Frame: Weeks 8, 9, 10, 11, 12, 13, and 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Percentage of participants
  Week 9 | 4.5 | 0.45 | 2.8
  Week 10 | 10.2 | 6.19 | 5.05
  Week 11 | 13.3 | 10.6 | 8.72
  Week 12 | 16.9 | 15.5 | 10.1
  Week 13 | 18.2 | 18.6 | 15.6
  Week 14 | 23.1 | 22.1 | 15.1
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.5279, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.37, 95% CI 2-sided [0.51 to 3.68]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 2]; Test type: Superiority or Other; p = 0.0141, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.13, 95% CI 2-sided [0.02 to 0.94]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 3]; Test type: Superiority or Other; p = 0.0484, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.92, 95% CI 2-sided [0.99 to 3.72]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 4]; Test type: Superiority or Other; p = 0.5813, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.23, 95% CI 2-sided [0.60 to 2.50]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 5]; Test type: Superiority or Other; p = 0.1236, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.51, 95% CI 2-sided [0.90 to 2.54]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 6]; Test type: Superiority or Other; p = 0.4998, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.21, 95% CI 2-sided [0.70 to 2.10]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.0365, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.64, 95% CI 2-sided [1.03 to 2.61]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 8]; Test type: Superiority or Other; p = 0.0822, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.52, 95% CI 2-sided [0.95 to 2.43]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 9]; Test type: Superiority or Other; p = 0.4049, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.19, 95% CI 2-sided [0.79 to 1.78]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; p = 0.2951, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.23, 95% CI 2-sided [0.84 to 1.80]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0248, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.53, 95% CI 2-sided [1.06 to 2.20]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.0326, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.51, 95% CI 2-sided [1.03 to 2.21]

20. Secondary Outcome: Percentage of Participants With a MADRS Response During Phase B Relative to the End of Phase A (Week 8 Visit) for the Efficacy Sample Per Final Protocol
Description: as for outcome 19
Time Frame: Weeks 8, 9, 10, 11, 12, 13, and 14
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Percentage of participants
  Week 9 | 3.37 | 0.48 | 3.02
  Week 10 | 7.58 | 6.1 | 4.93
  Week 11 | 13.3 | 11.3 | 8.37
  Week 12 | 16.6 | 16.4 | 10.3
  Week 13 | 18 | 19.2 | 14.3
  Week 14 | 23.2 | 23 | 14.3
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.7993, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.87, 95% CI 2-sided [0.30 to 2.55]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; p = 0.0118, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.11, 95% CI 2-sided [0.01 to 0.93]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 3]; Test type: Superiority or Other; p = 0.2825, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.50, 95% CI 2-sided [0.71 to 3.16]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.6375, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.20, 95% CI 2-sided [0.58 to 2.50]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 5]; Test type: Superiority or Other; p = 0.0923, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.62, 95% CI 2-sided [0.92 to 2.82]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 6]; Test type: Superiority or Other; p = 0.3812, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.29, 95% CI 2-sided [0.73 to 2.30]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 7]; Test type: Superiority or Other; p = 0.0464, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.63, 95% CI 2-sided [1.00 to 2.65]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 8]; Test type: Superiority or Other; p = 0.0490, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.62, 95% CI 2-sided [1.00 to 2.64]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 9]; Test type: Superiority or Other; p = 0.2124, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.32, 95% CI 2-sided [0.85 to 2.06]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 10]; Test type: Superiority or Other; p = 0.1078, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.41, 95% CI 2-sided [0.93 to 2.14]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0094, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.69, 95% CI 2-sided [1.14 to 2.50]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.0162, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.65, 95% CI 2-sided [1.09 to 2.50]

21. Secondary Outcome: Percentage of Participants With a MADRS Remission During Phase B Relative to the End of Phase A (Week 8) for the Efficacy Sample Set
Description: MADRS remission was defined as a < or equal to 10 and > or equal to 50% reduction in MADRS Total Score from end of Phase A (Week 8). The MADRS was utilized as an efficacy assessment of a participant's level of depression. The MADRS consisted of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS total score were to be unevaluable if less than 8 of the 10 items were recorded. If 8 or 9 of the 10 items were recorded, the MADRS total score was the mean of the recorded items multiplied by 10 and then rounded of to the first decimal place. The MADRS Total Score is the sum of ratings for all 10 items. The possible total scores are from 0 to 60, with higher values indicating worse outcome.
Time Frame: Weeks 8, 9, 10, 11, 12, 13 and 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 222 | 221 | 214
Percentage of participants
  Week 9 | 3.15 | 0.45 | 2.8
  Week 10 | 4 | 2.65 | 4.13
  Week 11 | 8.44 | 6.19 | 5.5
  Week 12 | 11.1 | 8.85 | 5.96
  Week 13 | 10.7 | 12.8 | 9.17
  Week 14 | 15.1 | 13.7 | 11.9
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.9498, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of remission rate = 1.03, 95% CI 2-sided [0.37 to 2.90]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 2]; Test type: Superiority or Other; p = 0.0141, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.13, 95% CI 2-sided [0.02 to 0.94]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 3]; Test type: Superiority or Other; p = 0.8609, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.93, 95% CI 2-sided [0.40 to 2.17]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 4]; Test type: Superiority or Other; p = 0.2846, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.59, 95% CI 2-sided [0.22 to 1.54]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 5]; Test type: Superiority or Other; p = 0.2480, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.50, 95% CI 2-sided [0.75 to 2.99]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 6]; Test type: Superiority or Other; p = 0.7513, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.13, 95% CI 2-sided [0.54 to 2.37]
Statistical Analysis 7: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.0554, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.82, 95% CI 2-sided [0.99 to 3.35]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 8]; Test type: Superiority or Other; p = 0.2409, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.48, 95% CI 2-sided [0.76 to 2.87]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 9]; Test type: Superiority or Other; p = 0.5538, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.18, 95% CI 2-sided [0.69 to 2.02]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; p = 0.1743, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.44, 95% CI 2-sided [0.85 to 2.41]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.2843, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.30, 95% CI 2-sided [0.81 to 2.07]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.4640, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.19, 95% CI 2-sided [0.74 to 1.92]

22. Secondary Outcome: Percentage of Participants With a MADRS Remission During Phase B Relative to the End of Phase A (Week 8) for the Efficacy Sample Per Final Protocol
Description: as for outcome 21
Time Frame: Weeks 8, 9, 10, 11, 12, 13 and 14
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Percentage of participants
  Week 9 | 1.92 | 0.48 | 3.02
  Week 10 | 2.37 | 2.82 | 3.94
  Week 11 | 8.06 | 6.57 | 5.42
  Week 12 | 10.4 | 9.39 | 6.4
  Week 13 | 9.95 | 13.1 | 8.37
  Week 14 | 14.7 | 14.1 | 10.8
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.3867, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.60, 95% CI 2-sided [0.18 to 1.97]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; p = 0.0118, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.11, 95% CI 2-sided [0.01 to 0.93]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 3]; Test type: Superiority or Other; p = 0.3200, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.59, 95% CI 2-sided [0.21 to 1.66]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.3266, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 0.60, 95% CI 2-sided [0.23 to 1.62]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 11 All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.3027, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.47, 95% CI 2-sided [0.70 to 3.10]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; Statistical analysis 2 at Week 11 All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.6960, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.17, 95% CI 2-sided [0.54 to 2.52]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; Statistical analysis 1 at Week 12 All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3. The LOCF method was used to impute missing data; Test type: Superiority or Other; p = 0.1368, Cochran-Mantel-Haenszel — CMH general association test controlling for trial site; Ratio of response rate = 1.62, 95% CI 2-sided [0.86 to 3.07]
Statistical Analysis 8: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 8]; Test type: Superiority or Other; p = 0.2387, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.48, 95% CI 2-sided [0.76 to 2.89]
Statistical Analysis 9: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 9]; Test type: Superiority or Other; p = 0.4498, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.26, 95% CI 2-sided [0.69 to 2.28]
Statistical Analysis 10: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 10]; Test type: Superiority or Other; p = 0.1009, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.60, 95% CI 2-sided [0.91 to 2.82]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1499, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.45, 95% CI 2-sided [0.87 to 2.41]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.3012, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.31, 95% CI 2-sided [0.78 to 2.18]

23. Secondary Outcome: Percentage of Participants With a CGI-I Response During Phase B Relative to the End of Phase A (Week 8 Visit) for the Efficacy Sample Set
Description: A CGI-I response was defined as a CGI-I score of 1 (very much improved) or 2 (much improved).
Time Frame: Weeks 8, 9, 10, 11, 12, 13 and 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 225 | 226 | 218
Percentage of participants
  Week 9 | 9.46 | 10.4 | 6.54
  Week 10 | 23.6 | 23 | 13.3
  Week 11 | 28.4 | 30.1 | 21.6
  Week 12 | 35.1 | 38.1 | 29.4
  Week 13 | 40 | 43.4 | 28.9
  Week 14 | 41.8 | 47.8 | 36.7
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.2873, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.41, 95% CI 2-sided [0.75 to 2.65]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 2]; Test type: Superiority or Other; p = 0.2677, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.37, 95% CI 2-sided [0.79 to 2.36]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 3]; Test type: Superiority or Other; p = 0.0031, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.80, 95% CI 2-sided [1.21 to 2.68]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 4]; Test type: Superiority or Other; p = 0.0066, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.70, 95% CI 2-sided [1.15 to 2.50]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 5]; Test type: Superiority or Other; p = 0.0665, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.34, 95% CI 2-sided [0.98 to 1.83]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 6]; Test type: Superiority or Other; p = 0.0250, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.41, 95% CI 2-sided [1.05 to 1.91]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.2224, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.18, 95% CI 2-sided [0.90 to 1.54]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 8]; Test type: Superiority or Other; p = 0.0369, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.31, 95% CI 2-sided [1.01 to 1.68]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 9]; Test type: Superiority or Other; p = 0.0179, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.36, 95% CI 2-sided [1.05 to 1.75]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.49, 95% CI 2-sided [1.17 to 1.89]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.3249, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.12, 95% CI 2-sided [0.89 to 1.41]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.0122, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.33, 95% CI 2-sided [1.06 to 1.66]

24. Secondary Outcome: Percentage of Participants With a CGI-I Response During Phase B Relative to the End of Phase A (Week 8 Visit) for the Efficacy Sample Per Final Protocol
Description: A CGI-I response was defined as a CGI-I score of 1 (very much improved) or 2 (much improved).
Time Frame: Weeks, 8, 9, 10, 11, 12, 13, and 14
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole (1mg) + ADT | Brexpiprazole (3mg) + ADT | Placebo + ADT
Number analyzed (Participants) | 211 | 213 | 203
Percentage of participants
  Week 9 | 7.69 | 9.52 | 5.53
  Week 10 | 21.8 | 23 | 12.3
  Week 11 | 27.5 | 30 | 19.7
  Week 12 | 34.1 | 38 | 27.6
  Week 13 | 38.9 | 44.1 | 27.1
  Week 14 | 41.2 | 48.4 | 34
Statistical Analysis 1: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.5836, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.22, 95% CI 2-sided [0.60 to 2.49]
Statistical Analysis 2: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; p = 0.3792, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.31, 95% CI 2-sided [0.73 to 2.37]
Statistical Analysis 3: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 3]; Test type: Superiority or Other; p = 0.0101, Ratio of response rate; CMH general association test controlling for trial site; Ratio of response rate = 1.77, 95% CI 2-sided [1.14 to 2.74]
Statistical Analysis 4: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.0065, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.75, 95% CI 2-sided [1.17 to 2.63]
Statistical Analysis 5: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 5]; Test type: Superiority or Other; p = 0.0526, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.41, 95% CI 2-sided [1.00 to 1.99]
Statistical Analysis 6: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 6]; Test type: Superiority or Other; p = 0.0156, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.51, 95% CI 2-sided [1.08 to 2.11]
Statistical Analysis 7: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 7]; Test type: Superiority or Other; p = 0.1689, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.22, 95% CI 2-sided [0.92 to 1.63]
Statistical Analysis 8: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 8]; Test type: Superiority or Other; p = 0.0231, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.37, 95% CI 2-sided [1.04 to 1.80]
Statistical Analysis 9: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 9]; Test type: Superiority or Other; p = 0.0175, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.40, 95% CI 2-sided [1.06 to 1.84]
Statistical Analysis 10: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 18, analysis 10]; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.59, 95% CI 2-sided [1.22 to 2.07]
Statistical Analysis 11: Comparison: Brexpiprazole (1mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.1396, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.21, 95% CI 2-sided [0.94 to 1.55]
Statistical Analysis 12: Comparison: Brexpiprazole (3mg) + ADT vs Placebo + ADT; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.0016, Cochran-Mantel-Haenszel; CMH general association test controlling for trial site; Ratio of response rate = 1.46, 95% CI 2-sided [1.15 to 1.86]

ADVERSE EVENTS:
Time Frame: AEs were captured from randomization to double-blind treatment at Week 8 to Follow-up 30 (+ 2) days after last dose of study medication.
Description: Safety sample comprised of randomized participants in Phase B who received at least one dose of double-blind trial medication. Participants were excluded only if there was evidence that the participant did not take trial medication. If a participant was dispensed trial medication and is lost to follow-up that participant was considered exposed.
Arm/Group | Brexpiprazole (1mg + ADT) | Brexpiprazole (3mg + ADT) | Placebo + ADT
Serious Adverse Events (participants affected / at risk) | 1/226 | 1/229 | 0/220
Other Adverse Events (participants affected / at risk) | 63/226 | 72/229 | 29/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (1mg + ADT) (N=226) | Brexpiprazole (3mg + ADT) (N=229) | Placebo + ADT (N=220)
Pneumonia (Infections and infestations) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (1mg + ADT) (N=226) | Brexpiprazole (3mg + ADT) (N=229) | Placebo + ADT (N=220)
Nasopharyngitis (Infections and infestations) | 15 | 7 | 4
Weight increased (Investigations) | 15 | 13 | 2
Akathisia (Nervous system disorders) | 10 | 31 | 5
Headache (Nervous system disorders) | 21 | 14 | 17
Somnolence (Nervous system disorders) | 9 | 13 | 1
Tremor (Nervous system disorders) | 9 | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No